CLINICAL TRIAL: NCT01302275
Title: Oxcarbazepine for the Treatment of Chronic Peripheral Neuropathic Pain: Predictors of Response - a Randomised, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Oxcarbazepine for the Treatment of Chronic Peripheral Neuropathic Pain
Acronym: IMIOXC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Søren H. Sindrup (Other)
Collaborators: Danish Pain Research Center (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor-Investigator, Søren H. Sindrup, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMIOXC
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Polyneuropathy; Peripheral Nerve Injury; Postherpetic Neuralgia
Keywords: neuropathic pain; oxcarbazepine; pain mechanism
MeSH Terms: conditions — Polyneuropathies; Peripheral Nerve Injuries; Neuralgia, Postherpetic; Neuralgia | interventions — Oxcarbazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxcarbazepine (Experimental): Oxcarbazepine is gradually increased during 21 days from 300 mg x 1 daily to 2400 mg, and kept on that dose ( 2400 mg) for three weeks.
  Interventions: Drug: Oxcarbazepine
- placebo (Placebo Comparator)
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine — Oxcarbazepine capsules 300 mg is gradually increased from 300 mg/day to 2400 mg/day Placebo capsules increase from 1/day to 8/day
  Other Names: Trileptal

SUMMARY:
The purpose of this trial is to determine if the effect of oxcarbazepine on chronic peripheral nerve pain depends on the supposed mechanism of the pain, ie. if oxcarbazepine mainly relieve pain in patients with irritable nerves.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* definite or probable neuropathic pain
* diagnosis of polyneuropathy, postherpetic neuralgia or peripheral nerve inju
* pain duration > 3 months
* pain rating at baseline >= 4 point NRS
* Informed consent

Exclusion Criteria:

* other non-neuropathic pain condition
* allergy to oxcarbazepine
* renal or hepatic impairment
* epilepsy
* depression and other serious psychiatric disorders
* serious medical condition
* previous treatment for neuropathic that cannot be stopped
* pregnancy
* patients expected not to be able to comply with study protocol
* treatment with anticonvulsants, antidepressant or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Total pain rated on numeric rating scale | Measurements from week 6 of treatment period
  Pain is rated daily on 0-10 point numeric rating scales. From the daily ratings from week 6 of each treatment period a median value is determined and used for data analysis. The analysis will compare scores between treatments (oxcabazepine vs placebo) and treatment effects (placebo-oxcarbazepine) between groups irritable nociceptor vs non-irritable nociceptors and some other subgroups.

SECONDARY OUTCOMES:
Response defined as at least 50% reduction in pain score | Week 6 of each treatment period vs. baseline
  Response defined as 50% reduction in pain score (median value week 6 of treatment period compared to median value during baseline period). Repsonse rates for each treatment and each phenotype will be calculated
Neuropathic Pain Symptom Inventory | Week 6 of each treatment period
  Different pain dimensions as rated by Neuropathic Pain Symptom Inventory
Patient Global Impression of Change | Week 6 of each treatment period
Rating of evoked pain | Week 6 of each treatment period
  Rating on numeric rating scales of pain induced by stimulation with cold rollers, stiff von Frey hain and dynamic touch with rubber sponge
Sleep disturbance | Week 6 of each treatment period
  Numeric rating scale ratings of pain induced sleep disturbance, median value of ratings from week 6 of each treatment period
Quality of life | Week 6 of each treatment period
  Rating of quality of life with numeric rating scale
Use of escape medication | Week 6 of each treatment period
  Number of paracetamol 500 mg used during the last week of each treamtent period

CONTACTS AND LOCATIONS:
Overall Officials: Søren H Sindrup, MD, Principal Investigator — Department of Neurology, Odense University Hospital
Locations (2):
- Denmark (2):
  - Danish Pain Research Center, Aarhus University Hospital, Aarhus
  - Department of Neurology, Odense University Hospital, Odense